CLINICAL TRIAL: NCT02175849
Title: Contact Tracing by Social Network Analysis to Enhance Multi-Drug Resistant Tuberculosis Case Finding in Hanoi, Vietnam
Brief Title: Intensifying Multi-Drug Resistant Tuberculosis Contact Tracing by Social Network Analysis
Acronym: SNAP
Status: Completed | Type: Observational
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: National Tuberculosis Program, Vietnam (Unknown)
Responsible Party: Sponsor
Other Study IDs: 10TB
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2014-07

CONDITIONS: Tuberculosis Infection
Keywords: Multi-Drug Resistant Tuberculosis; Social Network Analysis
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum Gastric Aspirate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Drug resistant TB patients: Patients with rifampicin resistant TB or MDR-TB newly confirmed by drug susceptibility tests (DST)
- Contacts: Contacts of patients with newly detected rifampicin resistant TB or MDR-TB in households, schools, workplaces and other locations.

SUMMARY:
Tuberculosis burden in Vietnam increasing with contribution from low detection rates and increased drug resistance. There is a need to identify MDR-TB (MultiDrug Resistant Tuberculosis) among both notified TB cases and their contacts in the community. Traditional contact tracing often focuses on household contacts while strains of TB circulate in homes, schools, workplaces, and beyond. Social network Analysis (SNA) is a comprehensive approach which includes a set of persons and the connections among them used for analysis of structure of disease transmission.

In this study, SNA will be used to collect network data from 60 newly detected Rifampicin resistant TB patients including an expected 50 MDR-TB patients living in Hanoi, and to identify and test potential MDR-TB cases.

DETAILED DESCRIPTION:
The study will identify and recruit 60 newly detected Rifampicin resistant TB patients including an expected 50 MDR-TB patients living in Hanoi (index cases) who will undergo SNA of contacts and places they have stayed during 3 months preceding their TB diagnosis including residence, travel history, places of social aggregation in relation with their risk behaviour.

Patients will be interviewed to investigate contacts before the confirmation of MDR-TB (for early contact detection and minimize the risk of information lost due to patient default during treatment). Data analysis will focus on MDR-TB social networks using Cytoscape software.

After the first two enrolled Rifampicin resistant MDR-TB cases, social network data will be analyzed to identify close contacts, mutual contacts, mutual places and high risk locations. The Social Network Questionnaire (SNQ) will be contextualized to the Vietnamese setting and validated in a pilot study. Eligible contacts and locations will undergo MDR-TB screening.

Approximately 720 contacts will undergo active screening (on 2 occasions per individual: at the time of contact identification and 6 months later). Contacts will include household contacts, close contacts, mutual contacts and symptomatic individuals with significant exposure to the index case at mutual locations within a closed environment.

Contact screening will involve clinical assessment, chest X-ray and sputum or gastric aspirate collection for TB culture, molecular techniques and microbiological identification.

If contacts are screened and detected as having Rifampicin resistant TB, they will be invited to be included in SNA for further analysis.

The number of MDR-TB detected by SNA will determine whether transmission of MDR-TB not otherwise detected by routine contact investigation (only household contact tracing) is important. While traditional contact tracing practices in Vietnam mainly focus on household contacts to detect secondary cases of TB, this SNA is expected not only to identify secondary cases of MDR-TB within an extended catchment but to also identify the source cases of MDR-TB patients to " turn off the tap" of MDR-TB transmission. Moreover, the places identified as the sources of sustained transmission will be targeted for case finding along with appropriate resource allocation.

In this study analysis will focus on the costs of contact tracing with Social Network Questionnaires, the proportion of MDR-TB among eligible contacts by subgroup, the proportion of MDR-TB among Rifampicin resistant TB patients and the genotyping pattern of MDR -TB patients.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS: Newly detected rifampicin resistant TB or MDR-TB patients living in Hanoi for at least 3 months preceding a diagnosis made between 2013-2015.
* CONTACTS: During the 3 months before the patient's TB or MDR-TB diagnosis: all persons who spend an average of >4 hours per day in the same residence as the patient AND/OR any individual who has had frequent and prolonged contact with the patient AND/OR anyone who has spent time in a closed environment with an MDR-TB patient
* PATIENTS AND CONTACTS: All ages
* PATIENTS AND CONTACTS: Living in Hanoi during the study period.

Exclusion Criteria:

-PATIENTS AND CONTACTS: Lack of informed consent for participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly detected rifampicin resistant TB or MDR-TB and their contacts
Sampling Method: Non-Probability Sample
Enrollment: 596 (Actual)
Dates: Start 2013-12; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Yield of MDR-TB case detection through SNA | Six months
  The number of MDR-TB cases notified from contacts identified by SNA and who would not have been detected by routine screening.

SECONDARY OUTCOMES:
MDR-TB incidence among subgroups of contacts | Six months
  The proportion of MDR-TB among eligible contacts by subgroup (household contacts, close contacts, mutual contacts, eligible contacts from mutual places with closed environment).
MDR-TB incidence among rifampicin resistant TB cases | Six months
  Incidence of MDR-TB confirmed by drug susceptibility tests (DST) among rifampicin resistant TB patients.
MDR-TB genotype | Six months
  Consistency or difference between TB genotype of enrolled MDR-TB patients and contacts/secondary cases.
Cost-effectiveness ratio of SNA and passive case finding strategies | Six months
  The incremental cost-effectiveness ratio (ICERs) between SNA and passive case finding for one MDR-TB case detected (i.e, the cost of SNA minus the cost of passive case finding divided by the yield in terms of case detection of SNA minus the yield of passive CF)

CONTACTS AND LOCATIONS:
Overall Officials: Heiman F Wertheim, PhD, Principal Investigator — Oxford University Clinical Research Unit - Hanoi
Locations (1):
- National Lung Hospital, Hanoi, Vietnam

REFERENCES:
- See also: Oxford University Clinical Research Unit — http://www.oucru.org